CLINICAL TRIAL: NCT00089076
Title: Phase I/II Study of Anti-CTLA-4 Monoclonal Antibody (MDX-010) in B-cell Non-Hodgkin's Lymphoma
Brief Title: MDX-010 in Treating Patients With Recurrent or Refractory Lymphoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02784; NCI-2012-02784 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC0312 (Other: Mayo Clinic); 6359 (Other: CTEP); P30CA015083 (NIH); U01CA069912 (NIH)
Record Dates: First submitted 2004-08-04; First posted 2004-08-05 (Estimated); Results first posted 2012-10-19 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2012-12

CONDITIONS: Adult Grade III Lymphomatoid Granulomatosis; B-cell Chronic Lymphocytic Leukemia; Cutaneous B-cell Non-Hodgkin Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Intraocular Lymphoma; Nodal Marginal Zone B-cell Lymphoma; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Refractory Hairy Cell Leukemia; Small Intestine Lymphoma; Splenic Marginal Zone Lymphoma; Testicular Lymphoma; Waldenström Macroglobulinemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Intraocular Lymphoma; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Hairy Cell; Waldenstrom Macroglobulinemia | interventions — Ipilimumab; CTLA-4 Antigen

ARMS (1):
- Treatment (ipilimumab) (Experimental): PHASE I: Patients receive MDX-010 IV over 90 minutes on day 1. Treatment repeats every 28 days for a total of 4 courses in the absence of disease progression or unacceptable toxicity.
  Cohorts of 6 patients from each group receive escalating doses of MDX-010 until the MTD is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.
  PHASE II: Patients receive MDX-010 as in phase I at the MTD.
  Interventions: Biological: ipilimumab; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: ipilimumab — Given IV
  Other Names: anti-cytotoxic T-lymphocyte-associated antigen-4 monoclonal antibody; MDX-010; MDX-CTLA-4; monoclonal antibody CTLA-4
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Biological therapies, such as MDX-010, work in different ways to stimulate the immune system and stop cancer cells from growing. This phase I/II trial is studying the side effects and best dose of MDX-010 and to see how well it works in treating patients with recurrent or refractory B-cell non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To characterize the safety profile of MDX-010 (ipilimumab) monoclonal antibody and identify a tolerable immunologically active dose level in B cell lymphoma patients.

II. To evaluate the clinical response rate in B cell lymphoma patients treated with MDX-010.

SECONDARY OBJECTIVES:

I. To evaluate the phenotype and function of memory T cells before and after treatment with MDX-010 by:

* Quantitation and phenotypic characterization of peripheral blood and tumor infiltrating T-cells, including cluster of differentiation (CD)4+CD25+ regulatory T cells.
* Measurement of tumor-specific T cells in peripheral blood lymphocytes.
* Measuring proliferation of memory T cells in response to recall antigens (tetanus toxoid and keyhole limpet hemocyanin [KLH]).

II. Measurement of anti-tumor antibodies in serum pre- and post-therapy. III. To evaluate the time to progression. IV. To evaluate the duration of response to treatment with MDX-010.

OUTLINE: This is a multicenter, open-label, phase I, dose-escalation study followed by a phase II study. Patients are grouped according to prior treatment with a vaccine therapy for lymphoma (yes vs no).

PHASE I: Patients receive anti-cytotoxic T-lymphocyte-associated antigen-4 monoclonal antibody (MDX-010) IV over 90 minutes on day 1. Treatment repeats every 28 days for a total of 4 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 6 patients from each group receive escalating doses of MDX-010 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

PHASE II: Patients receive MDX-010 as in phase I at the MTD.

Patients are followed at 1 and 4 months and then every 6 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologic proof of recurring or residual follicular B-cell non-Hodgkin's lymphoma (grade I or II), by Revised European American Lymphoma Classification (REAL) or World Health Organization (WHO) classifications which has relapsed or persisted after 3 or fewer conventional therapies, including chemotherapy or monoclonal antibody therapy; note: all patients with previously treated B-cell lymphomas of any histology with the exception of small lymphocytic lymphoma/chronic lymphocytic leukemia (CLL) are eligible
* Tumor measurable by computed tomography (CT) scans (at least one pathologic node measuring 2.0 x 2.0 cm, or 2 nodes measuring > 1.5 x 1.5 cm after collection of tumor for immunologic analyses)
* At least one prior treatment regimen but no more than 3 prior chemotherapy regimens; patients previously treated with monoclonal antibodies or radiotherapy to a single site will be eligible; these therapies will be considered prior treatment regimens but will not be considered as prior chemotherapy; tumor vaccines will not be counted as prior therapies, as all such agents are investigational
* Absolute neutrophil count (ANC) >= 1000/uL
* Platelets (PLT) >= 75,000/uL
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) =< 3 x upper limit or normal (ULN)
* Creatinine =< 1.5 x ULN
* Hemoglobin >= 8 g/dL
* Ability to provide informed consent
* Willingness to return to the Mayo Clinic Rochester or the University of California, Los Angeles for follow up
* Life expectancy >= 24 weeks
* Willingness to provide all biologic specimens as required by the protocol

Exclusion Criteria:

* Known standard therapy for the patient's disease that is potentially curative or definitely capable of extending life expectancy
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 2, 3, or 4
* Any uncontrolled infection, hepatitis C virus (HCV)+ (unless HCV ribonucleic acid [RNA]-negative by polymerase chain reaction [PCR]) or hepatitis B surface antigen (HBsAg)+, or human immunodeficiency virus (HIV) positive patients or patients with known immune deficiency states
* Previous MDX-010 therapy regardless of interval since last treatment
* Prior treatment with fludarabine or 2-chlorodeoxyadenosine =< 12 months prior to registration
* Failure to fully recover from acute, reversible effects of prior chemotherapy regardless of interval since last treatment
* New York Heart Association classification III or IV or a history of angina pectoris requiring active treatment
* Clinical evidence of central nervous system involvement by lymphoma
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception (condoms, diaphragm, birth control pills, injections, intrauterine device [IUD], or abstinence, etc.)
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational (utilized for a non-Food and Drug Administration [FDA]-approved indication and in the context of a research investigation)
* Diagnosis of small lymphocytic lymphoma/chronic lymphocytic leukemia (CLL)
* Any requirement for concurrent steroid therapy, including use of inhaled steroids for asthma
* History of autoimmune disease requiring systemic therapy with immunosuppressive drugs, including but not limited to rheumatoid arthritis, inflammatory bowel disease, systemic lupus erythematosus, multiple sclerosis, or psoriasis
* Antinuclear antibody (ANA) titer or rheumatoid factor titer > 3x institutional ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2004-06; Primary Completion 2008-07 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Ansell, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 2 medical clinics in the United States between August
  > 2004 and September 2007.
Pre-assignment Details: This was a phase I/II trial. A total of 18 participants were accrued, all to the phase I portion. This trial was terminated due to study design during the phase I; therefore, the phase II portion will never open. No results from the phase II portion are available.
Groups:
- MDX-010: Patients receive anti-cytotoxic T-lymphocyte-associated antigen-4 monoclonal antibody (MDX-010) IV over 90 minutes on day 1. Treatment repeats every 28 days for a total of 4 courses in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | MDX-010
Started | 18
Completed | 8
Not Completed | 10
Not completed — Alternate Therapy | 1
Not completed — Withdrawal by Subject | 2
Not completed — Progression | 7

BASELINE CHARACTERISTICS:
Arm/Group | MDX-010
Number analyzed (Participants) | 18
Age, Continuous [Median (Full Range); unit: years] | 56 [37 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 18
Disease Histology [Number; unit: participants]
  Follicular grade 1 lymphoma | 9
  Follicular grade 2 lymphoma | 5
  Diffuse large B-cell lymphoma | 3
  Mantle cell lymphoma | 1
Number of prior treatments [Median (Full Range); unit: Treatments] | 2 [1 to 4]
Dose Level [Number; unit: participants]
  3 mg/kg first dose, then 1 mg/kg monthly x 3 doses | 12
  3 mg/kg monthly x 4 doses | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Overall Confirmed Responses(Complete Response or Partial Response)
Description: Confirmed response is at least a 50% decrease in the sum of the products of the greatest diameters (SPD) of the six largest dominant nodes or nodal masses and no increase in the size of other nodes, liver, or spleen and splenic and hepatic nodules must regress by at least 50% in the SPD and no new sites of disease.
Time Frame: From registration to month 7
Measure: Number; unit: participants
Arm/Group | MDX-010
Number analyzed (Participants) | 18
participants | 2

2. Secondary Outcome: Time to Progression (Phase 2)
Description: The time to progression is defined as the time from registration to the time of progression. Those who die will be considered to have had disease progression unless documented evidence clearly indicates no progression has occurred. The distribution of time to progression will be estimated using the method of Kaplan-Meier.
Time Frame: From registration to progression (up to 2 years)
Population: No participants proceeded to Phase 2 for evaluation.
Arm/Group | MDX-010
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall Survival (Phase 2)
Description: The overall survival or survival time is defined as the time from registration to death due to any cause. The distribution of overall survival will be estimated using the method of Kaplan-Meier.
Time Frame: From registration to death (up to 2 years)
Population: No participants proceeded to Phase 2 for evaluation.
Arm/Group | MDX-010
Number analyzed (Participants) | 0

4. Secondary Outcome: Duration of Response (Phase 2)
Description: Duration of response will be calculated from the documentation of confirmed response until the date of progression in the subset of patients who respond.
Time Frame: From response to progression (up to 2 years)
Population: No participants proceeded to Phase 2 for evaluation.
Arm/Group | MDX-010
Number analyzed (Participants) | 0

5. Secondary Outcome: Mean Change in % of CD3+CD4+ for Marker HLA-DR+
Description: Flow cytometric analysis of T-cell surface markers before and 1 month after initiation therapy
Time Frame: Before treatment to 1 month after therapy initiation
Population: The analysis population contains patients that had peripheral blood available for analysis from before and 1 month after initiating therapy along with being able to conduct the analysis on the marker. This resulted in the number of participants analyzed being less than the enrolled participants.
Measure: Mean (Standard Error); unit: percentage of change of CD3+CD4+
Arm/Group | MDX-010
Number analyzed (Participants) | 14
percentage of change of CD3+CD4+ | 1.8 (1.2)

6. Secondary Outcome: Mean Change in % of CD3+CD4- for Marker HLA-DR+
Description: Flow cytometric analysis of T-cell surface markers before and 1 month after initiation therapy
Time Frame: Before treatment to 1 month after therapy initiation
Population: as for outcome 5
Measure: Mean (Standard Error); unit: percentage of change of CD3+CD4-
Arm/Group | MDX-010
Number analyzed (Participants) | 14
percentage of change of CD3+CD4- | 1.9 (2.0)

7. Secondary Outcome: Mean Change in % of CD3+CD4+ for Marker CD45RO+
Description: Flow cytometric analysis of T-cell surface markers before and 1 month after initiation therapy
Time Frame: Before treatment to 1 month after therapy initiation
Population: as for outcome 5
Measure: Mean (Standard Error); unit: percentage of change of CD3+CD4+
Arm/Group | MDX-010
Number analyzed (Participants) | 13
percentage of change of CD3+CD4+ | 5.0 (1.5)

8. Secondary Outcome: Mean Change in % of CD3+CD4- for the Marker CD45RO+
Description: Flow cytometric analysis of T-cell surface markers before and 1 month after initiation therapy
Time Frame: Before treatment to 1 month after therapy initiation
Population: as for outcome 5
Measure: Mean (Standard Error); unit: percentage of change of CD3+CD4-
Arm/Group | MDX-010
Number analyzed (Participants) | 13
percentage of change of CD3+CD4- | 2.8 (0.9)

ADVERSE EVENTS:
Arm/Group | MDX-010
Serious Adverse Events (participants affected / at risk) | 8/18
Other Adverse Events (participants affected / at risk) | 16/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MDX-010 (N=18)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Diarrhea-No Colostom (Gastrointestinal disorders) | 3 (3)
Fatigue (General disorders) | 1 (1)
Blood gonadotrophin abnormal (Investigations) | 1 (1)
Lymphopenia (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Weight loss (Investigations) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Facial nerve disorder (Nervous system disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MDX-010 (N=18)
Anemia (Blood and lymphatic system disorders) | 4 (7)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (3)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea-No Colostom (Gastrointestinal disorders) | 9 (11)
Dry mouth (Gastrointestinal disorders) | 1 (2)
Lip pain (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 3 (4)
Oral cavity Mucositis/stomatitis (functional/symptomatic) (Gastrointestinal disorders) | 1 (1)
Pain-Abdominal (Gastrointestinal disorders) | 6 (9)
Pain-Stomach (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Edema: Limb (General disorders) | 2 (2)
Fatigue (General disorders) | 12 (22)
Fever-No ANC (General disorders) | 2 (2)
Rigors (General disorders) | 1 (3)
Alkaline phosphatase (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 4 (5)
Creatinine (Investigations) | 1 (1)
Leukopenia (Investigations) | 4 (4)
Lymphopenia (Investigations) | 1 (1)
Neutropenia (Investigations) | 4 (5)
Platelet count decreased (Investigations) | 5 (9)
Weight loss (Investigations) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 4 (6)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (5)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (4)
Hypermatremia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 4 (6)
Impotence (Reproductive system and breast disorders) | 1 (3)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (5)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (5)
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 3 (6)
Sweating (Skin and subcutaneous tissue disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less